CLINICAL TRIAL: NCT06208293
Title: Opportunities for Suicide Prevention Integration Into Task-shifted Mental Health Interventions in Low-resourced Contexts
Brief Title: Suicide Prevention Integration Into Task-shifted Mental Health Interventions
Acronym: KPZ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000030402; K01MH125142 (NIH)
Record Dates: First submitted 2024-01-04; First posted 2024-01-17 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Suicide; Suicide Prevention; Suicidal Ideation
MeSH Terms: conditions — Suicide; Suicide Prevention; Suicidal Ideation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KPZ Program (KPZ) (Experimental): Participants in this group will receive the KPZ program in addition to EUC. This group will receive the culturally adapted suicide prevention package (KPZ) of services delivered by trained Peers. The KPZ package includes a culturally adapted approach to a co-designed safety plan. The assigned Peers will provide safety planning and Brief Contact Follow-Up. Contact follow up sessions will occur at the household level. A Peer will be assigned an eligible mother and visit her within no less than 48 hours of enrollment. The first session will be delivered within two days of detection, and follow up contacts conducted by a trained Peer at 24 hours, every two days (for one week), weekly (for 1 month), and monthly (for 5 months), totaling 13 KPZ sessions in all. Contact assesses how the participant is coping, if the safety plan is helpful, adjustments to the safety plan, assessment of the suicide ideation and depression, and providing basic motivational interviewing and referral as needed.
  Interventions: Behavioral: KPZ Program (KPZ); Behavioral: Enhanced Usual Care (EUC)
- Enhanced Usual Care (EUC) (Active Comparator): Participants in this group will receive usual care enhanced by Lady Health Workers (LHWs) trained in WHO Mental Health Gap Action Programme (mhGAP) that will link at-risk women with the primary care facility based medical officer. The LHWs will follow the mhGAP protocol for imminent or low risk of suicide including ensuring the participant is safe, removing or reducing means, assigning a family member to ensure safety (if appropriate), providing psychoeducation, and referring and accompanying the individual to their primary care health center where a mhGAP trained doctor is staffed to resume care or make a referral to specialized care. Additionally, all women and healthcare workers are provided a 24 hour hotline number (hosted by a Pakistani based mental health organization called Taskeen) and are briefed on exactly what will happen if participant calls.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: KPZ Program (KPZ) — The KPZ package includes a culturally adapted approach to a co-designed safety plan. The assigned Peers will provide safety planning and Brief Contact Follow-Up. Contact follow up sessions will occur at the household level.
  Arms: KPZ Program (KPZ)
Behavioral: Enhanced Usual Care (EUC) — Participants receive usual care enhanced by Lady Health Workers (LHWs) trained in WHO Mental Health Gap Action Programme (mhGAP) that will link at-risk women with the primary care facility based medical officer. The LHWs will follow the mhGAP protocol for imminent or low risk of suicide including ensuring the participant is safe, removing or reducing means, assigning a family member to ensure safety (if appropriate), providing psychoeducation, and referring and accompanying the individual to their primary care health center where a mhGAP trained doctor is staffed to resume care or make a referral to specialized care. Additionally, all women and healthcare workers are provided a 24 hour hotline number (hosted by a Pakistani based mental health organization called Taskeen) and are briefed on exactly what will happen if participant calls.

SUMMARY:
Investigators will conduct a pilot clinical trial to assess the feasibility and acceptability of implementing a Suicide Prevention Package (SuPP) within an existing task-shifted depression intervention in rural Pakistan. This pilot research lays the groundwork for a future project to scale a package for multi-level suicide prevention strategies that can be integrated into community based mental health programs, particularly targeting individuals living in low-resourced settings. As the model is designed to be easily adapted and integrated, investigators anticipate the findings will be valuable for all researchers looking to improve population health and mental health services in disadvantaged settings.

DETAILED DESCRIPTION:
The proposed research will (1) examine the epidemiology and health impacts of recurrent suicidal ideation on mothers over time, (2) characterize key features of suicidal ideation and finalize intervention package components within the study context, and (3) conduct a pilot clinical trial to assess the feasibility and acceptability of implementing a Suicide Prevention Package (SuPP) within an existing task-shifted depression intervention in rural Pakistan. This pilot research lays the groundwork for a future project to scale a package for multi-level suicide prevention strategies that can be integrated into community based mental health programs, particularly targeting individuals living in low-resourced settings. As the model is designed to be easily adapted and integrated, we anticipate the findings will be valuable for all researchers looking to improve population health and mental health services in disadvantaged settings. The focus of this registration is the pilot clinical trial.

A stratified cluster randomized controlled trial design, with 6 village clusters allocated in a 1:1 ratio to the intervention and control arms will be used. The stratification will be level of the Union Council (which is the smallest district administrative unit) and include Sihala and Shah Allah Ditta. While a village cluster (VC) will be the unit of randomization. Each VC will have 900-1400 population of women of reproductive age based within two to three contiguous catchment areas of the government employed community health workers called Lady Health Workers (LHWs). The reason for choosing village cluster as the unit of randomization is to minimize contamination/spillage between trial participants as the intervention will be delivered within community-based households. The intervention (KPZ) and control (EUC) village clusters will be geographically separated and the chance of intervention cluster participants regularly meeting control cluster participants will be negligible.

ELIGIBILITY:
Inclusion Criteria for trial participants receiving the intervention:

* Speak Urdu fluently
* Be actively receiving care from a clinician
* Have access to a mobile phone
* Intending to reside in the study area for the entire duration of the follow up (approx. six months)
* Has a child 3 years or under or is pregnant

Exclusion Criteria for trial participants receiving the intervention:

* Women requiring immediate inpatient care for any reason (medical or psychiatric)
* Women who do not speak and/or comprehend Urdu language

Inclusion Criteria for Peers and health system stakeholders:

* Speak Urdu fluently
* Be older than 18 at the time of recruitment
* Have access to a mobile phone
* Intending to reside in the study area for the entire duration of the follow up (approx. six months)

Exclusion Criteria for Peers and health system stakeholders:

* Women with untreated suicidality
* Women who do not speak and/or comprehend Urdu language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Mean score Beck's Scale for Suicidal Ideation (BSI) | baseline, 3 months and 6 months
  Suicide ideation severity measured with BSI. BSI is a 19-item self-report instrument for detecting and measuring the current intensity of the patients' specific attitudes, behaviors, and plans to commit suicide during the past week. The first 19 items consist of three options graded are on a 3-point scale ranging from 0 to 2. These items are then summed to yield a total score, which ranges from 0 to 38. Higher scores indicate more higher severity of suicide ideation.
Presence of any suicidal behaviors measured by the Columbia Suicide Severity Rating Scale (CSSRS) | baseline, 3 months and 6 months
  Suicidal behaviors and attempts measured with the CSSRS. The CSSRS asks about self-reported suicide attempt, aborted attempt, and interrupted attempt with "yes" or "no" questions. Any positive responses to these behaviors will be qualitatively coded as 'yes'. Behaviors are assessed at baseline as the past month and at 3 months and 6 months from the time of the previous assessment (e.g., past 3 months).
Percent eligible participants who consent | 6 months
  Percent eligible participants who agreed to participate
Percent of consented participants who started intervention | 6 months
  Percent consented participants who started intervention
Percent of participants who completed KPZ safety card | 6 months
  Percent of participants enrolled who completed KPZ safety card
Percent of participants who completed one brief contact follow up session | 6 months
  Percent of participants who completed one brief contact follow up session
Percent of participants who dropped out of KPZ intervention | 3 months and 6 months
  Percent of participants who dropped out of KPZ intervention
Median number of sessions completed | 6 months
  Median number of sessions completed by participants
Percent participants who completed all follow up measures | 6 months
  Percent participants who completed all follow up measures
Percent missing measure items per participant | 6 months
  Percent of missing measure items per participant

SECONDARY OUTCOMES:
Mean score on sub-scales of the Feasibility Acceptability and Appropriateness Measures of implementation (AIM/IAM). | 6 months
  All 3 scales are 4-items to assess core implementation outcomes of implementer perceptions of the KPZ intervention. FIM assesses if the intervention is feasible, possible, and easy, AIM assesses the implementation outcome of acceptability where respondents indicate their approval, find it appealing, express liking, and welcome the intervention strategy, providing valuable insights into the overall acceptability of the implemented approach. IAM measures appropriateness as an implementation outcome measuring if the intervention seems fitting, seems suitable, seems applicable, and seems like a good match. Responses for all scales use a 5-point ordinal likert scale, ranging from 1=completely disagree to 5=completely agree.
Mean score Knowledge, Attitudes, Self-efficacy, and practice of suicide prevention | 6 months
  The KAC is a 30-item questionnaire developed from our formative co-design research that assesses implementing agent (e.g., Peer) implementation domains of confidence (11 items), attitudes (acceptability, appropriateness, perceived benefit) (13 items), and knowledge (6 items) in implementing the elements of KPZ with the mother directly and within her social milieu (e.g., family engagement). The questionnaire assesses implementer understanding of their roles, confidence in identifying mothers at risk for suicide, and attitudes toward discussing and addressing suicide. Items are responded to with a 4-item Likert scale with responses ranging from 'none of the time' to 'all of the time'. The scale will be summed per sub-domain with a range of 0-39 for attitudes, 0-33 for confidence, and 0-18 for knowledge. Higher scores indicate more confidence, more positive attitudes, and more knowledge of KPZ intervention components and suicide myths.
Mean score Patient Health Questionnaire - 9 item (PHQ-9) | baseline, 3 months and 6 months
  Depression measured with PHQ-9. PHQ-9 is a 9-item validated questionnaire. Each item asks about the frequency of specific depressive symptoms experienced over the past two weeks. The response options are scored from 0 to 3, indicating "not at all" to "nearly every day." The item scores are summed with total score on the PHQ-9 ranges from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
Mean score Generalized Anxiety Disorder - 7 item (GAD-7) | baseline, 3 months and 6 months
  Anxiety measured with GAD-7, a 7 item self report instrument that measures anxiety Items are scored on a 4-point scale, ranging from "not at all (0)" to "nearly everyday (3)". Item scores are summed with a total score ranging from 0 to 21: 0-4 Minimal anxiety; 5-9 Mild anxiety; 10-14 Moderate anxiety; 15-21 Severe anxiety.
Mean score Multidimensional Scale of Perceived Social Support (MSPSS) | baseline, 3 months and 6 months
  The MSPSS is a 12 item questionnaire intended to measure the extent to which an individual perceives social support from Significant Others, Family and Friends. Each item is scored from 1 = Very Strongly Disagree, to 7 = very strongly agree). Total Scale: Sum across all 12 items, then divide by 12. Total score range from 1 to 7. Higher scores indicate more perceived social support.
Mean score Maternal Suicide Cognitions Scale | baseline, 3 months and 6 months
  Maternal Suicide Cognitions Scale (developed from formative interviews with 20 women with a history of suicidal behavior or clinical practice with suicidal women and 3 focus group discussions with Pakistani clinicians to identify inductively defined mechanisms of suicidality) includes presence of the following characteristics hypothesized to be on the pathway to suicidality including : loneliness, abandonment, helplessness, hopelessness, burdensomeness, anger, patience and other concepts rated on a 3-point likert scale. Item scores are summed. Scores range from 16 to 48 with higher scores indicated more risk cognitions.
Qualitative Interviews | 6 months
  Qualitative Interviews with trial participants, implementing agents (e.g., Peers and their supervisors), and health system stakeholders will elicit feasibility, acceptability, and perceived mechanisms of change. They will also inquire about adaptations (what, when, where, etc), familial, social and political factors that impacted KPZ implementation and engagement, and recommendations for changes for the future implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley K Hagaman, PhD MPH, Principal Investigator — Yale School of Public Health
Locations (1):
- Islamabad Capital Territory, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
What data that will be shared:
  Data associated with the trial will be deposited at ICPSR (Inter-university Consortium for Political and Social Research) which is an NIH-funded repository. Submitted data will conform with relevant data and terminology standards. The ICPSR website can be found here https://www.icpsr.umich.edu/web/pages/
  Who will have access to the data:
  Data will be deposited and made available through ICPSR which is an NIH-funded repository, and that these data will be shared with investigators requesting data working under an institution with a Federal Wide Assurance (FWA) and could be used for secondary study purposes such as meta analyses.
Supporting Information: Study Protocol
Time Frame: The data will become available as soon as possible but no later than within two years of the completion of the funded project period for the parent award or upon acceptance of the data for publication, whichever is earlier.
Access Criteria: Outcome data will be deposited in the ICPSR repository as soon as possible but no later than within two years of the completion of the funded project period for the parent award or upon acceptance of the data for publication, whichever is earlier.
  Investigators will identify where the data will be available and how to access the data in any publications and presentations that we author or co-author about these data, as well as acknowledge the repository and funding source in any publications and presentations. ICPSR has policies and procedures in place that will provide data access to qualified researchers, fully consistent with NIH data sharing policies and applicable laws and regulations.